CLINICAL TRIAL: NCT05778591
Title: Low-dose Buprenorphine as a Modulator of Social Motivation in Schizophrenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Anya Bershad, MD, PhD, Resident Physician, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB#23-000136
Record Dates: First submitted 2023-02-28; First posted 2023-03-21 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo, buprenorphine (Experimental): One group will receive placebo first, then buprenorphine (0.15mg).
  Interventions: Drug: Placebo; Drug: Buprenorphine 0.15 MG [Belbuca]
- Buprenorphine, placebo (Experimental): One group will receive buprenorphine (0.15mg) first, then placebo.
  Interventions: Drug: Placebo; Drug: Buprenorphine 0.15 MG [Belbuca]

INTERVENTIONS:
Drug: Placebo — Placebo.
Drug: Buprenorphine 0.15 MG [Belbuca] — Buprenorphine

SUMMARY:
Low social motivation is a significant symptom of schizophrenia and is a major cause of disability and suffering for many patients struggling with the illness. Social motivation refers to the drive to participate in or abstain from social activities. Many patients with schizophrenia evidence both decreased drive to seek positive social input (approach motivation) and heightened drive to avoid negative social input (avoidance motivation) compared to individuals without the illness. Despite the enormous burden of these deficits on patients, there are no medications that effectively treat impaired social motivation. Buprenorphine is an unusual drug that is used to treat opioid use disorder at higher doses and more recently, to treat depression and suicidality at lower doses. It is a unique opioid medication that has a compound action that gives it the potential to improve social motivation both by boosting approach motivation and by reducing avoidance motivation. The effects of low doses of buprenorphine have previously. been studied in healthy volunteers, showing that the drug enhances social motivation. These results in nonclinical volunteers suggest that buprenorphine may be a promising treatment for deficits in social motivation seen in some patients with schizophrenia. However, no previous studies have investigated the effects of buprenorphine on social motivation in this population. Here the effects of a low dose of buprenorphine (0.15mg) on social motivation in patients with schizophrenia (N=40) will be assessed. In this double-blind, cross-over, placebo-controlled study, participants will attend a 2-hour preparatory session and two 6-hour laboratory sessions, at which they will receive either placebo or buprenorphine. During expected peak drug effect they will complete validated tasks assessing social motivation. It is expected that buprenorphine will increase approach motivation and decrease avoidance motivation as measured by an attention bias task. The results of this study will lay the foundation for the clinical use of buprenorphine as the first medication to treat social deficits in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-60
2. able to understand spoken English sufficiently to comprehend testing procedures
3. score below the mean of participants screened previously screened on the Lubben Social Network Scale
4. DSM-5 diagnosis of schizophrenia
5. clinical stability (i.e., no inpatient hospitalizations for six months prior to enrollment, no changes in medication in for 6 months prior to enrollment, no current positive symptoms greater than moderate)

c) no history of IQ less than 70 or developmental disability, based on medical history d) no current use of opioid medication e) no clinically significant neurological disease (e.g., epilepsy), cardiovascular condition (e.g. cardiac arrhythmia), or respiratory condition (e.g., asthma) based on medical history

1. no history of serious head injury (i.e., loss of consciousness longer than 1 hour, neuropsychological sequelae, cognitive rehabilitation treatment after head injury) based on medical history
2. no substance or alcohol use disorder in the past six months, or history of opioid use disorder
3. no sedatives, benzodiazepines within 24 hours of testing
4. no positive urine toxicology screen or visible intoxication on the day of assessment
5. no women who are pregnant or think that they might be pregnant, based on self-report and urine test

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Attention bias | 90 minutes after drug administration
  Number of gazes toward each stimulus type on the attention bias task.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No